CLINICAL TRIAL: NCT06213948
Title: Elucidating Mechanisms That Underlie Symptomatology of Functional Dyspepsia Using Novel Imaging Technique of SPECT/CT, MRI, High-Resolution Manometry and Biomarkers; and the Therapeutic Validation of Elucidated Mechanisms Using Neuromodulator Compounds
Brief Title: Elucidating Mechanisms That Underlie the Symptomatology of Functional Dyspepsia Using Novel Techniques and Its Therapeutic Validation Using Neuromodulators
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Ministry of Higher Education, Malaysia (Other)
Responsible Party: Principal Investigator, Nashrulhaq Tagiling, MSc, PhD student, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: USM/JEPeM/20120624
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Functional Disorder of Stomach; Healthy
Keywords: Functional dyspepsia; Gastric accommodation; Gastric emptying; Micro inflammation
MeSH Terms: interventions — Mirtazapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy (Experimental)
  Interventions: Drug: Mirtazapine 15 MG
- Functional Dyspepsia (Experimental)
  Interventions: Drug: Mirtazapine 15 MG

INTERVENTIONS:
Drug: Mirtazapine 15 MG — Mirtazapine
  * Commercial name: Remeron® SolTab
  * Pharmaceutical form: film-coated tablets (15 mg)

SUMMARY:
The goal of this study is to investigate the mechanisms of impaired gastric accommodation and emptying, dysfunctional duodenum, and micro-inflammation using novel imaging techniques of SPECT/CT, gastric emptying scintigraphy, MRI, high-resolution manometry, and inflammatory biomarkers, as well as to validate these mechanisms using a therapeutic trial of neuromodulator (mirtazapine) in functional dyspepsia (FD) and health. The main objective[s] it aims to answer are:

* to investigate impaired gastric accommodation through SPECT/CT imaging and high-resolution manometry findings of the stomach fundus.
* to investigate impaired gastric emptying through gastric emptying scintigraphy
* to investigate for a dysfunctional duodenum through MRI imaging of the duodenum.
* to investigate micro-inflammation through SPECT/CT standard uptake value (SUV), inflammatory biomarkers (eosinophils, mast cells, IL-6, IL-10) and mucosal barrier marker (E-cadherin).
* to investigate if a therapeutic trial of a neuromodulator agent, mirtazapine, ameliorates symptoms of FD through improvement in impaired gastric accommodation.

For objectives 1-4, FD patients and healthy volunteers will be consecutively recruited, and all will undergo SPECT/CT, MRI, high-resolution manometry and biomarkers, and data acquired from these tests will be analyzed. For objective 5, the enrolled participants who did all baseline tests/markers are given mirtazapine for four weeks, and all tests/markers, except biomarkers and MRI, are repeated at the end of the trial

ELIGIBILITY:
Inclusion Criteria (Healthy):

* Age 18 and above, up to 65 years old
* No current GI symptoms (as assessed by history taking during screening and based on the investigators' collective judgement)
* No previous GI illness (as determined by clinically significant findings from medical history taking and vital signs)
* No chronic medical illness e.g., chronic neurological, cardiovascular, pulmonary, endoscirne and hematological disorders, as well as psychiatric disorders

Exclusion Criteria (Healthy):

* BMI of less than 18.50 and more than 29.99
* Had undergone any abdominal surgery except appendicectomy, tubal ligation, or Caesarean section
* Females that are pregnant, expecting to become pregnant during the study period, or breastfeeding
* Aversion to test meals
* Use of medications that may alter gastrointestinal function and motility
* Contraindication for MRI examination e.g., cardiac pacemaker, ferromagnetic implants, claustrophobia

Inclusion Criteria (FD patients):

* Age 18 and above, up to 65 years old
* Satisfy the diagnosis of FD as per Rome IV criteria
* Absence of organic disorders that explain dyspepsia in patients such as autoimmune disease, inflammatory disease or brain trauma
* No other chronic medical illnesses (including chronic neurological, cardiovascular, pulmonary, endocrine and hematological disorders) and psychiatric disorders

Exclusion Criteria (FD patients):

* Positive Helicobacter pylori test
* Presence of esophagitis, gastric atrophy, heartburn as predominant symptom, history of peptic ulcer or major abdominal surgery
* Medications that potentially affects gastrointestinal motility or sensitivity (eg: acid suppressant, prokinetics, corticosteroids, NSAIDs and analgesics apart from paracetamol)
* Aversion to test meals
* Recent trauma to the abdomen
* Patients on antipsychotic or antidepressant in the last 6 weeks
* Contraindication for MRI examination e.g., cardiac pacemaker, ferromagnetic implants, claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastric volume (fasting and postprandial) | Fasting, 10-min. postprandial
  SPECT/CT volumetry
Gastric emptying profile (4 hours) | Immediately after test meal ingestion, up to 4 hours postprandial
  Gastric emptying scintigraphy
Intragastric pressure | Fasting, up to 30-min. postprandial after reaching maximum tolerated volume
  High-resolution manometry

SECONDARY OUTCOMES:
Satiation | Fasting, up to 30-min. postprandial after reaching maximum tolerated volume
  Satiation scale
Upper gastrointestinal symptoms | Fasting, up to 30-min. postprandial after reaching maximum tolerated volume
  Visual analog scale

OTHER OUTCOMES:
Standardized Uptake Value (stomach) | Fasting and 10-min. postprandial
  SPECT/CT quantitative imaging

CONTACTS AND LOCATIONS:
Overall Officials: Nashrulhaq Tagiling, MSc, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing has yet to be discussed thoroughly with co-investigators.